CLINICAL TRIAL: NCT01026246
Title: Phase I, Double-Blinded, Placebo-Controlled Dosage-Escalation Study of the Safety and Immunogenicity of EBA-175 RII-NG Malaria Vaccine Administered Intramuscularly in Semi-immune Adults
Brief Title: EBA-175 RII-NG Malaria Vaccine Administered Intramuscularly in Semi-immune Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 08-0009
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2012-05

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Ghana, malaria, vaccine, Plasmodium falciparum
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Group B: 20 mcg EBA-175 + 500 mcg aluminum phosphate adjuvant (Experimental): 18 subjects to receive 20 mcg EBA-175 + 500 mcg aluminum phosphate adjuvant; 2 subjects to receive placebo.
  Interventions: Drug: Placebo; Biological: EBA-175 RII-NG Malaria Vaccine
- Group A: 5 mcg EBA-175 + 500 mcg aluminum phosphate adjuvant (Experimental): 18 subjects to receive 5 mcg EBA-175 + 500 mcg aluminum phosphate adjuvant; 2 subjects to receive placebo.
  Interventions: Drug: Placebo; Biological: EBA-175 RII-NG Malaria Vaccine
- Group C: 80 mcg EBA-175 + 500 mcg aluminum phosphate adjuvant (Experimental): 18 subjects to receive 80 mcg EBA-175 + 500 mcg aluminum phosphate adjuvant; 2 subjects to receive placebo.
  Interventions: Drug: Placebo; Biological: EBA-175 RII-NG Malaria Vaccine

INTERVENTIONS:
Drug: Placebo — The placebo used will be normal saline (0.9 percent NaCl).
Biological: EBA-175 RII-NG Malaria Vaccine — EBA-175 RII-NG malaria vaccine is supplied as a white, translucent, cloudy, nonparticulate liquid suspension in single-dose clear glass vials pre-mixed with Adju-Phos aluminum phosphate adjuvant. Each 2-mL vial of EBA-175 RII-NG vaccine contains: 0.7 mL (0.5 mL per dose) EBA-175 RII-NG, at the required dose concentration, 5 percent sucrose, 1.0 mg/mL (0.5 mg/0.5 mL per dose) aluminum as aluminum phosphate adjuvant, sodium phosphate buffer (10 mM sodium phosphate and 150 mM sodium chloride), and no preservative.

SUMMARY:
Malaria is caused by a germ that people get from the bites of some mosquitoes. It kills over 2 million people each year. Many of the drugs used to treat malaria do not work as well as they used to and researchers are exploring other vaccines to prevent malaria. The purpose of this study is to learn if the vaccine, called EBA-175 RII-NG, is safe and if it strengthens the body's defenses against malaria. Participants will include 60 healthy adults, ages 18-40, recruited from Accra, Ghana. Several dosages of the vaccine will be tested for safety. The lowest dosages of the vaccine will be tested before the next higher dose is tested. There will be two groups for each dose, one group will receive the vaccine and the other group will receive a placebo (salt water solution). Participants may be involved in study related procedures for up to 398 days.

DETAILED DESCRIPTION:
Malaria accounts for 500 million febrile illnesses and more than a million deaths annually. The disease burden is heaviest in economically developing countries where it is estimated that up to 5 percent of the gross domestic product of sub-Saharan countries is consumed by the direct and indirect health costs of malaria. Researchers propose to conduct a Phase I dosage-escalating study to assess the safety and immunogenicity of 3 different dosages of erythrocyte-binding antigen 175 kDA region II-nonglycosylated (EBA-175 RII-NG) recombinant Plasmodium falciparum (Pf) vaccine adjuvanted with Adju-Phos (aluminum phosphate adjuvant): 5, 20, and 80 micrograms (mcg), given in 3 doses at 0, 1, and 6 months by intramuscular (IM) injection to healthy young adults in a malaria endemic area (semi-immune adults). One dose of vaccine will be given at each time point. The primary objective is to assess the safety and reactogenicity (tolerability) of ascending dosages of EBA-175 RII-NG vaccine among healthy subjects given in 3 IM doses at 0, 1 and 6 months. The secondary objective is to evaluate the immunogenicity of the EBA-175 RII-NG vaccine by measuring anti-EBA-175 RII-NG antibodies using enzyme-linked immunosorbent assay (ELISA), inhibition of Plasmodium falciparum growth in vitro, and inhibition of binding of EBA-175 RII-NG to red blood cells (RBCs). Participants will include 60 malaria semi-immune healthy subjects between the ages of 18 and 40 years, males and females, recruited from Accra, Ghana. Subjects will be randomized to receive 3 doses of the vaccine or saline placebo by the intramuscular route in a 9:1 ratio at 0, 1 and 6 months. The safety and immunogenicity of ascending dosages of the vaccine will be assessed. Eighteen subjects will receive vaccine at each of the following dosage levels: 5, 20, and 80 mcg. Two subjects will receive placebo for each dosage level. Dosage escalation will proceed only after review of the 2-week safety data of the 2 initial doses of the prior dosage level.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and healthy non-pregnant and non breastfeeding females between the ages of 18 and 40 years.
* Females of childbearing potential must agree to practice adequate contraception through out the study and for 3 months after the third vaccination (including abstinence; hormonal contraception; condoms with spermicidal agents); males with female partners of childbearing age must agree to use condoms or other birth control.
* Good health as determined by screening medical history, physical examination (PE), and routine laboratory assessments.
* Willingness to comply with protocol requirements.
* Ability to provide informed consent before any protocol procedures are performed.
* Availability for follow-up for 12 months after the first immunization dose.

Exclusion Criteria:

* Regular use of medications other than vitamins and contraceptives.
* Current or recent (within the last 4 weeks prior to vaccination) treatment with parenteral, inhaled, or oral corticosteroids (intranasal steroids are acceptable), or other immunosuppressive agents, or chemotherapy.
* History of splenectomy.
* Abnormal screening laboratory values. Any abnormal screening value for any screening test, will exclude the subject from the study. An exception to this rule is the glucose measurement. Random plasma glucose will be measured on all subjects during the screening visit. Values higher than 110 mg/dl will be confirmed by a repeat fasting glucose measurement.
* History of or current medical, occupational, social or family problems as a result of alcohol or illicit drug use by the volunteer.
* History of moderate to severe mental illness, as defined by symptoms interfering with social or occupational function or suicidal thoughts/attempts.
* History of receiving blood or blood products (such as blood transfusion, platelet transfusion, immunoglobulins, hyperimmune serum) in the previous 6 months.
* Vaccination with a live vaccine within the past 30 days or with a non-replicating, inactivated, or subunit vaccine within the last 14 days.
* Known hypersensitivity to components of the vaccine [Erythrocyte-Binding Antigen 175 kDa Region II-Nonglycosylated (EBA-175 RII-NG), sucrose, or aluminum adjuvant].
* History of acute or chronic medical conditions including, but not limited to, disorders of the liver, kidney, lung, heart, or nervous system, or other metabolic and autoimmune/inflammatory conditions, sickle cell disease.
* History of anaphylaxis or severe hypersensitivity reaction.
* Severe asthma, as defined by an emergency room visit or hospitalization within the last 12 months.
* Pregnant or breastfeeding women, or women unwilling to use effective contraception during the study period.
* Acute illness, including temperature > 37.8 degrees Celsius within one week prior to vaccination.
* Positive serology for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B surface antigen (HBsAg).
* Concurrent participation in other investigational protocols or receipt of an investigational product within the previous 30 days.
* Identification of any condition that, in the opinion of the investigator, would affect the ability of the subject to understand or comply with the study protocol or would jeopardize the safety or rights of a subject participating in the study.
* History of malignancy, including hematologic and skin cancers, or known immunodeficiency syndrome.
* Pre-medication with analgesic or antipyretic in the 6 hours prior to vaccination, or planned medication with analgesic or antipyretic in the 24 hours following vaccination. This criterion should not preclude subjects receiving such medication after vaccination if the need arises.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing severe (Grade 3) solicited injection site reactions. | Within 14 days following vaccination.
Number of subjects experiencing severe solicited systemic reactions (Grade 3). | Within 14 days following vaccination.
Number of subjects experiencing severe (Grade 3) clinical laboratory values. | Within 14 days following vaccination.
Number of subjects spontaneously reporting adverse events considered associated with the vaccination that are severe (Grade 3). | Duration of study.
Serious adverse events considered associated with the vaccination. | Duration of study.

SECONDARY OUTCOMES:
Number of subjects experiencing a 4-fold increase in Anti-EBA-175 RII-NG antibody level (ELISA). | Days 14, 28, 42, 180 and 194 relative to baseline.
Relative binding inhibition of recombinant EBA-175 RII-NG to human red blood cells in vitro in the presence of serum from immunized individuals. | Days 0, 14, 28, 42, 180 and 194.
Anti-EBA-175 RII-NG antibody level by enzyme-linked immunosorbent assay (ELISA). | Days 0, 14, 28, 42, 180 and 194.
Relative growth inhibition of Plasmodium falciparum in human red blood cells cultured in vitro in the presence of serum from immunized individuals. | Days 0, 14, 28, 42, 180 and 194.

CONTACTS AND LOCATIONS:
Locations (1):
- Noguchi Memorial Institute for Medical Research - Immunology, Legon, Greater Accra Region, Ghana

REFERENCES:
- [Derived] Koram KA, Adu B, Ocran J, Karikari YS, Adu-Amankwah S, Ntiri M, Abuaku B, Dodoo D, Gyan B, Kronmann KC, Nkrumah F. Safety and Immunogenicity of EBA-175 RII-NG Malaria Vaccine Administered Intramuscularly in Semi-Immune Adults: A Phase 1, Double-Blinded Placebo Controlled Dosage Escalation Study. PLoS One. 2016 Sep 19;11(9):e0163066. doi: 10.1371/journal.pone.0163066. eCollection 2016. PMID 27644034